CLINICAL TRIAL: NCT04635917
Title: Effects of a Personalized Functional Food Diet on Cardiometabolic, Microbiome and Metabolomics Profiles in Minority Young Adults
Brief Title: Effects of a Personalized Diet on Cardiometabolic, Microbiome and Metabolomics Profiles in Minority Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jaapna Dhillon, Assistant Professor, Nutrition & Exercise Phys-MED, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022561; R00MD012815 (NIH)
Record Dates: First submitted 2020-10-26; First posted 2020-11-19 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Diet Intervention
Keywords: Personalized

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Personalized diet - Black adults (Experimental): Young Black adults in this group will receive tailored nutrition counseling from a dietitian. To facilitate meeting their dietary goals, participants will be provided with nuts, fruits, and vegetables.
  Interventions: Other: Personalized diet
- Personalized diet - White adults (Experimental): Young White adults in this group will receive tailored nutrition counseling from a dietitian. To facilitate meeting their dietary goals, participants will be provided with nuts, fruits, and vegetables.
  Interventions: Other: Personalized diet
- Conventional dietary advice- Black adults (Other): Young Black adults will receive non-personalized, conventional dietary advice based on the MyPlate guidelines.
  Interventions: Other: Conventional dietary advice
- Conventional dietary advice- White adults (Other): Young White adults will receive non-personalized, conventional dietary advice based on the MyPlate guidelines.
  Interventions: Other: Conventional dietary advice

INTERVENTIONS:
Other: Personalized diet — Participants in this group will receive tailored nutrition counseling from a dietitian. To facilitate meeting these dietary goals, participants will be provided with nuts, fruits, and vegetables.
  Other Names: PD
  Arms: Personalized diet - Black adults; Personalized diet - White adults
Other: Conventional dietary advice — Participants in the CD group will receive non-personalized, conventional dietary advice by a dietitian based on the MyPlate guidelines.
  Other Names: CD
  Arms: Conventional dietary advice- Black adults; Conventional dietary advice- White adults

SUMMARY:
The proposed study has two primary objectives i.e. to examine how improvements in diet quality via a personalized dietary intervention 1) benefit cardiometabolic outcomes in young Black adults differentially compared to non-Hispanic White adults, and 2) improve carbohydrate and lipid metabolism in relation to the gut microbiome.

DETAILED DESCRIPTION:
The study is an 8-wk randomized, controlled, parallel arm clinical trial in which participants (age: 18-35 years, BMI: 25-45 kg/m2, race/ethnicity: Black or White) will be block randomized to a personalized dietary intervention or to receive conventional dietary advice. Outcomes assessed will include metabolites involved in carbohydrate and lipid regulation, gut microbiome composition, and cardiometabolic biomarkers.

ELIGIBILITY:
Inclusion criteria:

* Age: 18-35 years of age
* BMI: 25-45 kg/m2
* Black including those of Hispanic ethnicity, and Non-Hispanic White individuals
* Willingness to consume nuts, fruits and vegetables
* Willing to comply with study protocol
* Consistent diet and activity patterns for 4 weeks
* Weight stable (≤5 kg change over the last 3 months) (Self-reported)
* Non-smoker >1 year or more

Exclusion Criteria:

* Allergies to fruits, vegetables, and nuts provided in the study
* Illicit drug use
* Recent start of medications that affect metabolism or appetite
* Antibiotics
* Coronary artery disease, peripheral artery disease, congestive heart failure, or dyslipidemia requiring drug therapy
* Uncontrolled hypertension and blood pressure ≥ 180/110 Diabetes
* Gastrointestinal disease and/or bariatric surgery
* HIV positivity
* Pregnant or lactating individuals

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Change in diet quality | Change over 8 weeks
  Healthy eating index score
Change in relative intensities of metabolites in blood | Change over 8 weeks
  Measured by untargeted metabolomics mass spectrometry
Change in stool microbiome profiles | Change over 8 weeks
  16s rRNA sequencing
Change in endothelial function | Change over 8 weeks
  Reactive hyperemia index
Matsuda index | Change over 8 weeks
  Assessed via a 2-hour oral glucose tolerance test
Change in lipid profile | Change over 8 weeks
  LDL, HDL, triglycerides, total cholesterol
Change in glucoregulation | Change over 8 weeks
  Fasting glucose concentrations
Change in insulinemic biomarker concentrations | Change over 8 weeks
  Fasting insulin and C-peptide concentrations
Change in blood pressure | Change over 8 weeks
  Diastolic and systolic blood pressure
Change in inflammatory markers | Change over 8 weeks
  MCP-1,IL6, IL10, TNFa, hs-CRP, and fibrinogen

SECONDARY OUTCOMES:
Body Mass | Every 2 weeks over the 8 week intervention
  Body mass will be measured in kg
Body Composition | Every 2 weeks over the 8 week intervention
  Fat mass, fat-free mass
Anthropometrics | Every 2 weeks over the 8 week intervention
  Waist circumference, hip circumference
24-hour appetite ratings | Every 4 weeks over the 8 week intervention
  Subjective ratings using visual analog scales
Physical activity | Every 4 weeks over the 8 week intervention
  Activity assessment using Actigraphs
Palatability rating of foods | Every 2 weeks over the 8 week intervention
  Hedonic general labelled magnitude scale (gLMS)
Acceptance rating of foods | Every 2 weeks over the 8 week intervention
  9-point food action rating scale

OTHER OUTCOMES:
Transcriptomics profiles | Baseline and at the end of the 8-week intervention
  Untargeted transcriptomics
Attention score | Change over 8 weeks
  d2 test of attention
Memory | Change over 8 weeks
  Word recall scores
Food environment perceptions | Baseline and at the end of the 8-week intervention
  Subjective and objective questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jaapna Dhillon, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported here after deidentification (ie; text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Data will be deposited in NIH supported data repositories.

DOCUMENTS (1):
  • Informed Consent Form (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT04635917/ICF_000.pdf